CLINICAL TRIAL: NCT05290987
Title: Efficacy of ADW S-100 Ionized Water Nasal Spray in Decreasing SARS-Cov-2 Viral Load in Adults With High Viral Excretion by Nasopharyngeal Swabbing. Randomized, Double-blind, Placebo-controlled, Parallel Group Study.
Brief Title: Efficacy of ADW S-100 Ionized Water Nasal Spray in Decreasing SARS-Cov-2 Viral Load.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of participants needed not reached (13/80)
Sponsor: P & B Group (Industry)
Collaborators: MediAxe CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-A01861-40
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Water S-100 ionized nasal spray (Experimental): 2 sprays in each nostril, 6 times a day during 8 days
  Interventions: Device: nasal spray
- Nasal spray with purified water (Placebo Comparator): 2 sprays in each nostril, 6 times a day during 8 days
  Interventions: Device: nasal spray

INTERVENTIONS:
Device: nasal spray — 2 sprays in each nostril, 6 times a day

SUMMARY:
A nasal spray based on Advanced Water S-100 ionized water would clean the nasal cavity, reduce the viscosity of the mucus and facilitate its elimination and the decongestion of the nose and the prevention of the seizure of the SARS-COV-2 to the epithelial cells of the nasal cavity In fact, a nasal spray based on Advanced Water S-100 ionized water would modify the electrostatic environment of all interactions ensuring this seizure. The negative ions (OH-) contained in Advanced Water S-100 compete with the negative ions of the heparan sulfate, which will destabilize this essential bond for the virus to enter the host cell. In addition, positively charged basic amino acids, in the presence of the basic pH of ADW S-100, will be neutralized by OH- ions which will prevent the formation of salt and hydrogen bridges mediating the formation of the protein S/ACE2 complex. The destabilization of all bonds governing the protein S/ACE2 association process will prevent the virus from entering cells and replicating.

The aim of this study is to evaluate whether the use of ADW S-100 ionized water nasal spray reduces the salivary and nasopharyngeal viral load during an 8-day follow-up of persons recently infected with SARS-Cov-2, and thus potentially decreases the risk of contamination of the entourage.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old
2. Informed consent
3. Beneficiaries of a social security plan
4. Vaccinated or unvaccinated against SARS-COV-2:

   * Vaccinated individuals have had a 3rd dose for at least one month, or have been infected with SARS-Cov-2 and have had 2 doses of vaccine for at least one month
   * Unvaccinated persons are naïve to previous SARS Cov 2 infection
5. Positive nasopharyngeal RT-PCR test for selection with a Ct viral load ≤ 23
6. Have a phone and internet connection to access the entry application

Exclusion Criteria:

1. The participant is related to any member of the study staff or has a close relationship or conflict of interest with the sponsor.
2. Known hypersensitivity or allergy to any component of the test product.
3. Contraindication to nasal spray
4. Insufficient vaccination: any incomplete vaccination schedule

   * either a 3rd dose within the last month
   * or SARS-Cov-2 infection with less than 2 vaccine doses or with 2 vaccine doses less than 1 month old.
5. Any condition, including COVID, that is likely to result in hospitalization during study participation.
6. Conditions that may result in hospitalization during study participation.
7. Known pregnancy or positive urine pregnancy test at D0 by the nurse, or current breastfeeding
8. Participation in an antiviral clinical trial or other trial using a medical device for disease prevention COVID 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
To determine whether, compared to placebo, ADW S-100 ionized water administered as a nasal spray more rapidly negatively affects the viral load of individuals infected with SARS-CoV-2 | 8 days
  % of participants negative at D4 (Ct≥35)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Bouvier, Dr, Principal Investigator — independent oto rhino laryngologist
Locations (1):
- Dr Bouvier's Office, Aix-en-Provence, France

IPD SHARING:
Plan to Share IPD: No
Trial prematurely stopped as recruitment interrupted with less than 10% participants included